CLINICAL TRIAL: NCT00721097
Title: Predictive Factors for Exacerbation Outcome in Severe Refractory Asthmatics
Acronym: EXPRESA
Status: Terminated | Type: Observational
Why Stopped: Number of included patients is sufficient.
Sponsor: Nantes University Hospital (Other)
Responsible Party: General Director, Nantes University Hospital
Other Study IDs: BRD 07/6-X
Record Dates: First submitted 2008-07-07; First posted 2008-07-23 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Asthma; Chronic Inflammatory Diseases
Keywords: Severe asthma; exacerbation; predictive factors; Severe
MeSH Terms: conditions — Asthma; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: spirometry, and blood taken — each month during one year

SUMMARY:
Asthma is a chronic inflammatory disease, affecting up to 10 % of the general population in developed countries. Corticosteroids are necessary to control symptoms, but induce adverse events sometimes intolerable. In severe asthma, which represent 5 to 10% of global asthma, corticosteroids frequently fail to prevent severe exacerbations, leading to emergency care, hospitalization and sometimes death. The aim of this study is to identify predictive factors specific for exacerbation outcome which will lead to a minor increase in treatment in order to prevent exacerbations, while minimizing drug adverse effects.

ELIGIBILITY:
Inclusion criteria :

* Male or female adults aged ≥ 18 years, who have signed an Inform Consent Form prior to initiation of any study-related procedure
* Patients with severe asthma with at least 2 exacerbations during the last 12 months that necessitated oral cortico-therapy or increase in oral cortico-therapy

Exclusion criteria :

* Pregnant or nursing women
* Patients with other chronic inflammatory lung disease
* Current smoker or a smoking history of 10 pack years or more

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe asthma
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Number of predictive factors for exacerbation outcome in severe asthmatics.

SECONDARY OUTCOMES:
Rate of predictive factors identified in the study, in order to prevent exacerbations.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine MAGNAN, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- nantes University Hospital, Nantes, Nantes, France